CLINICAL TRIAL: NCT05762276
Title: A Phase 1, First-in-Human, Dose Escalation Study to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacodynamics of VXX-401 in Healthy Adults
Brief Title: A Study to Investigate the Safety, Tolerability, Immunogenicity, and Pharmacodynamics of VXX-401 Administered IM in Adult Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vaxxinity, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VXX-401-101
Record Dates: First submitted 2023-02-20; First posted 2023-03-09 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cohorts A-D are blinded / Cohort E & F are open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- VXX-401 Cohort A (Experimental): VXX-401 100mcg administered by intramuscular (IM) injection at Week 0, Week 4, and Week 12
  Interventions: Drug: VXX-401
- VXX-401 Cohort B (Experimental): VXX-401 100mcg administered by intramuscular (IM) injection at Week 0, Week 4, Week 8 and Week 12
  Interventions: Drug: VXX-401
- VXX-401 Cohort C (Experimental): VXX-401 300mcg administered by intramuscular (IM) injection at Week 0, Week 4, and Week 12
  Interventions: Drug: VXX-401
- VXX-401 Cohort D (Experimental): VXX-401 300mcg administered by intramuscular (IM) injection at Week 0, Week 4, Week 8 and Week 12
  Interventions: Drug: VXX-401
- Placebo Cohort A and C (Placebo Comparator): Placebo administered by intramuscular (IM) injection at Week 0, Week 4, and Week 12
  Interventions: Biological: Placebo
- Placebo Cohort B and D (Placebo Comparator): Placebo administered by intramuscular (IM) injection at Week 0, Week 4, Week 8 and Week 12
  Interventions: Biological: Placebo
- VXX-401 Cohort E (Experimental): VXX-401 900mcg administered by intramuscular (IM) injection at Week 0. VXX-401 100 mcg administered by intramuscular (IM) injection at Week 4 and Week 12.
  Interventions: Drug: VXX-401
- VXX-401 Cohort F (Experimental): VXX-401 900mcg administered by intramuscular (IM) injection at Week 0. VXX-401 300 mcg administered by intramuscular (IM) injection at Week 4 and Week 12.
  Interventions: Drug: VXX-401

INTERVENTIONS:
Drug: VXX-401 — A synthetic PCSK9 peptide-based immunotherapy
  Arms: VXX-401 Cohort A; VXX-401 Cohort B; VXX-401 Cohort C; VXX-401 Cohort D; VXX-401 Cohort E; VXX-401 Cohort F
Biological: Placebo — Normal saline
  Arms: Placebo Cohort A and C; Placebo Cohort B and D

SUMMARY:
This first-in-human (FIH) study of VXX-401, an anti-PCSK9 peptide-based immunotherapeutic candidate, is designed to assess the safety, tolerability, immunogenicity, and pharmacodynamics (PD) of VXX-401 and to determine an optimal dose regimen for LDL-C lowering in subsequent clinical trials.

DETAILED DESCRIPTION:
This is multisite, multidose regimen, phase 1, first-in-human study of VXX-401, a synthetic peptide-based active immunotherapy candidate for preventing and treating hypercholesterolemia. The study will include Screening, Treatment, and Follow-up Periods. This study will enroll participants who are naïve to statin use. Each cohort from A to D is planned to randomize approximately 12 participants to receive doses of VXX-401 or placebo in a 3:1 ratio. Cohorts E and F will dose approximately 8 participants in each cohort to receive doses of VXX-401. No participants will be administered placebo in Cohorts E and F. It is planned to test up to 6 dose regimens of VXX-401, administered by IM injection into the deltoid muscle (and additionally in the thigh for the first dose in Cohorts E-F.). All eligible participants will receive a priming regimen at Week 0 (Baseline, Day 1), Week 4, and Week 12, in Cohorts A, C, E and F, and additionally at Week 8 in Cohorts B and D. The last dose administration will be at Week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 to 75 years old, inclusive, at time of informed consent.
2. LDL-C level = 2.59 mmol/L - 4.89mmol/L
3. Body mass index between 18 and 35 kg/m2, inclusive at Screening, and with a minimum weight of 50 kg.
4. Male participants and their partners of childbearing potential must commit to the use of highly effective contraceptives for the study duration and for at least 12 weeks after the last dose. Men must refrain from donating sperm during this same period.
5. Female participants must be of nonchildbearing potential, or, for women of childbearing potential, must be willing to practice at least one form of highly effective contraception throughout the duration of the study and for at least 24 weeks following the last dose. Female participants must refrain from donating reproductive tissue during this same period.

Exclusion Criteria:

1. Subjects considered high risk or very high risk for ASCVD and requiring immediate treatment with LLT according to the clinical judgement of the investigator.
2. History of confirmed anergy (i.e., not able to mount an immunological response) or history of immunization failure in the 5 years prior to the Screening Visit.
3. Presence of fever >38°C or other signs or symptoms of acute disease within 1 week before the Screening and/or Visit 1; Screening and/or Visit 1 may be rescheduled at the discretion of the Investigator but must occur within the 4-week window.
4. Known disturbance of coagulation or medication (see prohibited medications criterion below); bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
5. Triglycerides > 5.65 mmol/L
6. Has a history of clinically significant medical disorder or psychiatric conditions, which in the opinion of the investigator may compromise the participant's safety and ability to comply with study procedures or abide by study restrictions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-06-27 (Estimated); Study Completion 2024-06-27 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events | 30 weeks
  Safety and tolerability: rates of adverse events (AEs), medically attended adverse events (MAAEs), local (injection site) and systemic (generalized) reactions (i.e., reactogenicity), clinical laboratory assessments (e.g., chemistry, hematology, urinalysis, lipid profile), serum cytokine release, vital signs, physical examinations, and electrocardiograms (ECGs) through the end of the study.
Immunogenicity | Baseline to Week 16, 20, 24, and 30
  Immunogenicity will be measured by serum anti-PCSK9 antibody titers
Immunogenicity | Baseline to Week 16, 20, 24, and 30
  Seroconversion two-fold and four-fold from baseline
Determine optimal VXX-401 dose regimen | Baseline to Week 16, 20, 24, and 30
  Measured by serum anti-PCSK9 antibody titers

SECONDARY OUTCOMES:
Evaluation of low-density lipoprotein-cholesterol (LDL-C) reduction | Baseline to Week 16, 20, 24, and 30
  Percent change from baseline in serum LDL-C concentration

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Rumyantsev, Study Director — Vaxxinity, Inc.
Locations (5):
- Australia (5):
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Sutherland Shire Clinical Research, Miranda, New South Wales
  - Emeritus Research, Sydney, New South Wales
  - University of the Sunshine Coast (USC), Morayfield, Queensland
  - Emeritus Research, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No